CLINICAL TRIAL: NCT06684925
Title: Relationship Between Stability of Cervical Spine With Function and Grade Point Average in University Students
Brief Title: Stability and Function of Cervical Spine With Grade Point Average in University Students
Status: Active, not recruiting | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Assistant professor of physical therapy for neurology, Al-Ahliyya Amman University
Other Study IDs: 10566
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cervical Lesion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal disorders are some of the most prevalent health concerns, especially among students

DETAILED DESCRIPTION:
Stability of the cervical spine during head and cervical movements is an important component of cervical spine function .The deep neck flexor (DNF) (longus colli, longus capitis) muscles stabilize the neck and contribute to the control of head acceleration. Weakening of these muscles can lead to its coordination, activation, overload and poor support in the cervical structures. Further causes neck pain and altered neck position.

Studies conducted on patients with neck pain have also shown activation of these muscles and reduced resistance, associated disorders and headaches. Muscle resistance should be considered as a measure of neck function or injury.

University class, staying up late can be considered a risk factor for neck pain in students.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 20 to 25 years old
* Students have no health problems or complains

Exclusion Criteria:

* neck pain
* Cervical radiculopathy
* Fracture
* Previous back problems
* Students with low grade (GPA below 2)

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 124 students of both genders (42 males, 82 females) that agreed to participate, were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Hand Held Dynamometer | Two months
  was used to measure deep neck flexors isometric strength.
Neck disability index | Two months
  is a reliable, validated and clinically useful tool to measure disability due to neck pain. It is designed to measure "activity limitations" during activities of daily living (ADL) in patients with neck pain.It is divided into 10 items, four related to participant symptoms (pain intensity, headache, concentration, and sleep), four related to ADL (lifting things, working, driving a car, and having fun), and two related to personal care and reading. Each of the items is scored from zero to five points Disability was classified as: absent (total score between zero and 4 points); mild (total score between 5 and 14 points); moderate (total score between 15 and 24 points); severe (total score between 25 and 34 points); and complete (total score above 34 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Ahliyya Amman University, Amman, Jordan